CLINICAL TRIAL: NCT01821118
Title: A Phase 2, Randomized, Double Blind Placebo Controlled Trial To Evaluate The Safety, Tolerability, Pharmacokinetics And Efficacy Of Pf-04360365 (Ponezumab) In Adult Subjects With Probable Cerebral Amyloid Angiopathy
Brief Title: Study Evaluating the Safety,Tolerability and Efficacy of PF-04360365 in Adults With Probable Cerebral Amyloid Angiopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A9951024; 2013-001557-27 (EudraCT Number)
Record Dates: First submitted 2013-03-04; First posted 2013-03-29 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Cerebral Amyloid Angiopathy
Keywords: Cerebral amyloid angiopathy (CAA); cerebrovascular reactivity; functional MRI; randomized; double blind; safety; efficacy
MeSH Terms: conditions — Cerebral Amyloid Angiopathy | interventions — ponezumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: Ponezumab
- 2 (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Biological: Ponezumab — Infusion of Ponezumab (Day 1=10mg/kg; Day 30 and Day 60 dose = 7.5mg/kg) or placebo (saline); administered via infusion for a total infusion time of 20 minutes.
  Arms: 1
Other: placebo — placebo (saline)- given via infusion total infusion time of 20 minutes
  Arms: 2

SUMMARY:
Cerebral Amyloid Angiopathy (CAA) is a condition caused by the build-up of a protein called amyloid, predominantly Aβ40, within the walls of brain blood vessels, especially those blood vessels in the occipital lobe of the brain. Probable CAA may be defined as two or more hemorrhages in the brain cortex in individuals 55 years of age or older. This study will examine the study drug (PF-04360365) vs. placebo (saline) at 10 mg/kg - Day 1 and the maintenance dose of the study drug (PF-04360365) vs. placebo (saline) at 7.5mg/kg on Days 30 and 60. Subjects will be followed for 6 months after receiving the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with probable CAA using the Boston criteria; with no clinical cognitive impairment
* In general good health

Exclusion Criteria:

* Co-morbid diagnosis of clinically documented Alzheimer's disease or significant cognitive impairment
* Clinically significant syncope, epilepsy, head trauma or clinically significant unexplained loss of consciousness within the last 5 years
* Subject's body weight exceeding 100kg
* Women of childbearing potential.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (7):
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - MGH Stroke Research Center, Boston, Massachusetts
  - Boston Medical Center - Menino Pavilion, Boston, Massachusetts
  - Boston Medical Center - Shapiro Center, Boston, Massachusetts
  - Anthinoula A. Martinos Center for Biomedical Imaging, Charlestown, Massachusetts
  - Barnes Jewish Hospital, St Louis, Missouri
  - Columbia University, New York, New York
- Canada (2):
  - University of Calgary/Foothills Medical Centre, Calgary, Alberta
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- France (2):
  - CHRU de Lille - Hôpital Roger Salengro, Lille, NAP
  - CHRU de Lille, Lille, NAP
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands
- University College of London, London, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9951024&StudyName=Study%20Evaluating%20the%20Safety%2CTolerability%20and%20Efficacy%20of%20PF-04360365%20in%20Adults%20with%20Probable%20Cerebral%20Amyloid%20Angiopathy%20

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04360365: Participants received a loading dose of PF-04360365 10 milligrams (mg)/kilograms (kg) on Day 1, followed by PF-04360365 7.5 mg/kg on Days 30 and 60. PF-04360365 was administered via intravenous (IV) infusion over a period of 10-15 minutes (min) and dosing was based on participant weight.
- Placebo: Participants received a loading dose of placebo matching PF-04360365 10 mg/kg on Day 1, followed by placebo matching PF-04360365 7.5 mg/kg on Days 30 and 60. Placebo was also administered via IV infusion over a period of 10-15 min.
Period: Overall Study
Arm/Group | PF-04360365 | Placebo
Started | 24 | 12
Completed | 24 | 11
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants assigned to study treatment were included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04360365 | Placebo | Total
Number analyzed (Participants) | 24 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (6.8) | 65.0 (5.7) | 67.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 16 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 2 in Cerebrovascular Reactivity as Measured by the Slope (Amplitude Over Time to Peak) From Visual Task-evoked Functional Magnetic Resonance Imaging (fMRI)
Description: Blood Oxygen Level Dependant (BOLD) fMRI was performed at Screening (Baseline) and on Days 2 and 90. During each of these sessions, BOLD fMRI images were acquired in rapid succession as a flashing radial black and white checkerboard was presented alternately with a gray screen. This well established visual stimulus is known to produce a reliable increase in BOLD fMRI signal within the visual cortex region of the occipital lobe. The time course of the BOLD fMRI signal was used to assess the vascular reactivity. Imaging sites also acquired cerebral blood flow data using Arterial Spin Labeled (ASL) scans at Screening and on Days 2 and 90. A standard T1-weighted image was also acquired to aid image analysis. All efficacy scans were analyzed centrally. Geometric means are presented in the original scale and standard errors (SE) are presented in logarithmic (log e) scale.
Time Frame: Baseline, Day 2
Population: The full analysis set (FAS) consisted of all participants who received at least 1 post-dose efficacy measurement. n=number of evaluable participants for the specified region of interest (ROI) at Day 2.
Measure: Geometric Mean (Standard Error); unit: percent/second
Arm/Group | PF-04360365 | Placebo
Number analyzed (Participants) | 24 | 12
percent/second
  Region of interest (ROI) 1 (n=20, 11) | 0.954 (0.085) | 0.969 (0.073)
  ROI2 (n=23, 11) | 0.933 (0.050) | 0.999 (0.055)
Statistical Analysis 1: Comparison: PF-04360365 vs Placebo; ROI1: Analysis of the change from baseline in log(slope) was carried out using a Bayesian linear model (ANCOVA). Treatment was a fixed effect within the model and the log(slope) at baseline was included as a covariate; Test type: Superiority or Other; Geometric Mean Ratio = 0.984, 90% CI 2-sided [0.820 to 1.184], Standard Error of Mean 0.112 — SE of mean is presented in log e scale
Statistical Analysis 2: Comparison: PF-04360365 vs Placebo; ROI2: Analysis of the change from baseline in log(slope) was carried out using a Bayesian linear model (ANCOVA). Treatment was a fixed effect within the model and the log(slope) at baseline was included as a covariate; Test type: Superiority or Other; Geometric Mean Ratio = 0.934, 90% CI 2-sided [0.825 to 1.056], Standard Error of Mean 0.075 — SE of mean is presented in log e scale

2. Primary Outcome: Change From Baseline to Day 90 in Cerebrovascular Reactivity as Measured by the Slope (Amplitude Over Time to Peak) From Visual Task-evoked fMRI
Description: BOLD fMRI was performed at Screening (Baseline) and on Days 2 and 90. During each of these sessions, BOLD fMRI images were acquired in rapid succession as a flashing radial black and white checkerboard was presented alternately with a gray screen. This well established visual stimulus is known to produce a reliable increase in BOLD fMRI signal within the visual cortex region of the occipital lobe. The time course of the BOLD fMRI signal was used to assess the vascular reactivity. Imaging sites also acquired cerebral blood flow data using ASL scans at Screening and on Days 2 and 90. A standard T1-weighted image was also acquired to aid image analysis. All efficacy scans were analyzed centrally. Geometric means are presented in the original scale and SEs are presented in log e scale.
Time Frame: Baseline, Day 90
Population: The full analysis set (FAS) consisted of all participants who received at least 1 post-dose efficacy measurement. n=number of evaluable participants for the specified ROI at Day 90.
Measure: Geometric Mean (Standard Error); unit: percent/second
Arm/Group | PF-04360365 | Placebo
Number analyzed (Participants) | 24 | 12
percent/second
  ROI1 (n=20, 10) | 0.817 (0.064) | 0.958 (0.063)
  ROI2 (n=23, 10) | 0.857 (0.055) | 0.950 (0.060)
Statistical Analysis 1: Comparison: PF-04360365 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric Mean Ratio = 0.852, 90% CI 2-sided [0.735 to 0.989], Standard Error of Mean 0.091 — SE of mean is presented on log e scale
Statistical Analysis 2: Comparison: PF-04360365 vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Geometric Mean Ratio = 0.902, 90% CI 2-sided [0.788 to 1.031], Standard Error of Mean 0.082 — SE of mean presented on log e scale

3. Secondary Outcome: Change From Baseline to Day 2 and Day 90 in Cerebrovascular Reactivity as Measured by the Time to Peak From Visual Task-evoked fMRI
Description: as for outcome 2
Time Frame: Baseline, Day 2, Day 90
Population: The full analysis set (FAS) consisted of all participants who received at least 1 post-dose efficacy measurement. n=number of evaluable participants for the specified ROI at the specified day.
Measure: Geometric Mean (Standard Error); unit: seconds
Arm/Group | PF-04360365 | Placebo
Number analyzed (Participants) | 24 | 12
seconds
  ROI1, Day 2 (n=20, 11) | 1.012 (0.028) | 1.007 (0.037)
  ROI1, Day 90 (n=20, 10) | 1.065 (0.020) | 1.015 (0.030)
  ROI2, Day 2 (n=23, 11) | 1.008 (0.018) | 1.010 (0.026)
  ROI2, Day 90 (n=23, 10) | 1.039 (0.018) | 1.028 (0.026)
Statistical Analysis 1: Comparison: PF-04360365 vs Placebo; ROI1, Day 2: Analysis of the change from baseline in log(time to peak) was carried out using a Bayesian linear model (ANCOVA). Treatment was a fixed effect within the model and the log(time to peak) at baseline was included as a covariate; Test type: Superiority or Other; Geometric Mean Ratio = 1.005, 90% CI 2-sided [0.933 to 1.086], Standard Error of Mean 0.046 — SE of mean presented on log e scale
Statistical Analysis 2: Comparison: PF-04360365 vs Placebo; ROI1, Day 90: Analysis of the change from baseline in log(time to peak) was carried out using a Bayesian linear model (ANCOVA). Treatment was a fixed effect within the model and the log(time to peak) at baseline was included as a covariate; Test type: Superiority or Other; Geometric Mean Ratio = 1.049, 90% CI 2-sided [0.990 to 1.114], Standard Error of Mean 0.036 — SE of mean presented on log e scale
Statistical Analysis 3: Comparison: PF-04360365 vs Placebo; ROI2, Day 2: Analysis of the change from baseline in log(time to peak) was carried out using a Bayesian linear model (ANCOVA). Treatment was a fixed effect within the model and the log(time to peak) at baseline was included as a covariate; Test type: Superiority or Other; Geometric Mean Ratio = 0.998, 90% CI 2-sided [0.947 to 1.052], Standard Error of Mean 0.032 — SE of mean presented on log e scale
Statistical Analysis 4: Comparison: PF-04360365 vs Placebo; ROI2, Day 90: Analysis of the change from baseline in log(time to peak) was carried out using a Bayesian linear model (ANCOVA). Treatment was a fixed effect within the model and the log(time to peak) at baseline was included as a covariate; Test type: Superiority or Other; Geometric Mean Ratio = 1.010, 90% CI 2-sided [0.960 to 1.063], Standard Error of Mean 0.031 — SE of mean presented on log e scale

4. Secondary Outcome: Change From Baseline to Day 2 and Day 90 in Cerebrovascular Reactivity as Measured by the Amplitude From Visual Task-evoked fMRI
Description: BOLD fMRI was performed at Screening (Baseline) and on Days 2 and 90. During each of these sessions, BOLD fMRI images were acquired in rapid succession as a flashing radial black and white checkerboard was presented alternately with a gray screen. This well established visual stimulus is known to produce a reliable increase in BOLD fMRI signal within the visual cortex region of the occipital lobe. The time course of the BOLD fMRI signal was used to assess the vascular reactivity. Imaging sites also acquired cerebral blood flow data using ASL scans at Screening and on Days 2 and 90. A standard T1-weighted image was also acquired to aid image analysis. All efficacy scans were analyzed centrally. All values are presented in log e scale.
Time Frame: Baseline, Day 2, Day 90
Population: as for outcome 3
Measure: Least Squares Mean (90% Confidence Interval); unit: percent
Arm/Group | PF-04360365 | Placebo
Number analyzed (Participants) | 24 | 12
percent
  ROI1, Day 2 (n=20, 11) | -0.0381 (0.028) [-0.1655 to 0.0894] | -0.0983 (0.037) [-0.2715 to 0.0750]
  ROI1, Day 90 (n=20, 10) | -0.1389 (0.020) [-0.2513 to -0.0264] | -0.053 (0.030) [-0.2135 to 0.1075]
  ROI2, Day 2 (n=23, 11) | -0.0714 (0.018) [-0.1584 to 0.0156] | -0.0226 (0.026) [-0.1484 to 0.1033]
  ROI2, Day 90 (n=23, 10) | -0.1245 (0.018) [-0.2236 to -0.0254] | -0.0357 (0.026) [-0.1861 to 0.1146]
Statistical Analysis 1: Comparison: PF-04360365 vs Placebo; ROI1, Day 2: Analysis of the change from baseline in log(amplitude) was carried out using a linear model (ANCOVA). Treatment was a fixed effect within the model and the log(amplitude) at baseline was included as a covariate; Test type: Superiority or Other; Estimated Treatment Difference (log e) = 0.0602, 90% CI 2-sided [-0.1576 to 0.2781], Standard Error of Mean 0.1281
Statistical Analysis 2: Comparison: PF-04360365 vs Placebo; ROI1, Day 90: Analysis of the change from baseline in log(amplitude) was carried out using a linear model (ANCOVA). Treatment was a fixed effect within the model and the log(amplitude) at baseline was included as a covariate; Test type: Superiority or Other; Estimated Treatment Difference (log e) = -0.0859, 90% CI 2-sided [-0.2843 to 0.1124], Standard Error of Mean 0.1165
Statistical Analysis 3: Comparison: PF-04360365 vs Placebo; ROI2, Day 2: Analysis of the change from baseline in log(amplitude) was carried out using a linear model (ANCOVA). Treatment was a fixed effect within the model and the log(amplitude) at baseline was included as a covariate; Test type: Superiority or Other; Estimated Treatment Difference (log e) = -0.0488, 90% CI 2-sided [-0.2018 to 0.1042], Standard Error of Mean 0.0902
Statistical Analysis 4: Comparison: PF-04360365 vs Placebo; ROI2, Day 90: Analysis of the change from baseline in log(amplitude) was carried out using a linear model (ANCOVA). Treatment was a fixed effect within the model and the log(amplitude) at baseline was included as a covariate; Test type: Superiority or Other; Estimated Treatment Difference (log e) = -0.0888, 90% CI 2-sided [-0.2689 to 0.0914], Standard Error of Mean 0.1061

5. Secondary Outcome: Change From Baseline to Day 2 and Day 90 in Cerebrovascular Reactivity as Measured by the Time to Return to Baseline From Visual Task-evoked fMRI
Description: as for outcome 4
Time Frame: Baseline, Day 2, Day 90
Population: as for outcome 3
Measure: Least Squares Mean (90% Confidence Interval); unit: seconds
Arm/Group | PF-04360365 | Placebo
Number analyzed (Participants) | 24 | 12
seconds
  ROI1, Day 2 (n=20, 11) | 0.0245 (0.028) [-0.0155 to 0.0644] | -0.022 (0.037) [-0.0759 to 0.0319]
  ROI1, Day 90 (n=20, 10) | 0.0558 (0.020) [0.0182 to 0.0934] | -0.0179 (0.030) [-0.0711 to 0.0354]
  ROI2, Day 2 (n=23, 11) | 0.0045 (0.018) [-0.0280 to 0.0369] | -0.0174 (0.026) [-0.0643 to 0.0295]
  ROI2, Day 90 (n=23, 10) | 0.0275 (0.018) [-0.0040 to 0.0589] | 0.0158 (0.026) [-0.0322 to 0.0637]
Statistical Analysis 1: Comparison: PF-04360365 vs Placebo; ROI1, Day 2: Analysis of the change from baseline in log(time to return to baseline) was carried out using a linear model (ANCOVA). Treatment was a fixed effect within the model and the log(time to return to baseline) at baseline was included as a covariate; Test type: Superiority or Other; Estimated Treatment Difference (log e) = 0.0464, 90% CI 2-sided [-0.0207 to 0.1136], Standard Error of Mean 0.0395
Statistical Analysis 2: Comparison: PF-04360365 vs Placebo; ROI1, Day 90: Analysis of the change from baseline in log(time to return to baseline) was carried out using a linear model (ANCOVA). Treatment was a fixed effect within the model and the log(time to return to baseline) at baseline was included as a covariate; Test type: Superiority or Other; Estimated Treatment Difference (log e) = 0.0737, 90% CI 2-sided [0.0084 to 0.1390], Standard Error of Mean 0.0383
Statistical Analysis 3: Comparison: PF-04360365 vs Placebo; ROI2, Day 2: Analysis of the change from baseline in log(time to return to baseline) was carried out using a linear model (ANCOVA). Treatment was a fixed effect within the model and the log(time to return to baseline) at baseline was included as a covariate; Test type: Superiority or Other; Estimated Treatment Difference (log e) = 0.0219, 90% CI 2-sided [-0.0352 to 0.0790], Standard Error of Mean 0.0337
Statistical Analysis 4: Comparison: PF-04360365 vs Placebo; ROI2, Day 90: Analysis of the change from baseline in log(time to return to baseline) was carried out using a linear model (ANCOVA). Treatment was a fixed effect within the model and the log(time to return to baseline) at baseline was included as a covariate; Test type: Superiority or Other; Estimated Treatment Difference (log e) = 0.0117, 90% CI 2-sided [-0.0460 to 0.0694], Standard Error of Mean 0.034

6. Secondary Outcome: Change From Baseline in Concentration of Total Plasma Amyloid Beta (AB)
Description: Cerebral amyloid angiopathy (CAA) is caused by the progressive deposition of amyloid, predominantly AB40, within the walls of cerebral blood vessels with a predisposition for the vessels of the occipital lobe. As such, it is of interest to investigate the effect of PF-04360365 on AB concentrations. AB1-x and AB1-40 were investigated.
Time Frame: Baseline, 8 hours post dose on Day 1, Day 2, Day 30, 90 and 240
Population: All 36 participants who received study treatment were included in this pharmacodynamic analysis. n=number of participants with measurable AB at the specified time point.
Measure: Mean (Standard Deviation); unit: picograms (pg)/milliliter (mL)
Arm/Group | PF-04360365 | Placebo
Number analyzed (Participants) | 24 | 12
picograms (pg)/milliliter (mL)
  AB1-x, Day 1 (n=4, 3) | 4374.0 (420.62) | 5.3 (26.01)
  AB1-x, Day 2 (n=4, 3) | 13911.8 (3292.88) | -37.7 (29.02)
  AB1-x, Day 30 (n=4, 3) | 94468.5 (11946.21) | -48.3 (103.32)
  AB1-x, Day 90 (n=4, 2) | 111312.8 (24677.74) | -62.0 (141.42)
  AB1-x, Day 240 (n=4, 3) | 30495.8 (10931.16) | 13.0 (116.76)
  AB1-40, Day 1 (n=23, 11) | 4747.6 (1039.96) | -8.4 (30.08)
  AB1-40, Day 2 (n=23, 11) | 12845.2 (2887.91) | 0.5 (30.90)
  AB1-40, Day 30 (n=23, 10) | 68010.1 (17396.04) | -5.0 (46.81)
  AB1-40, Day 90 (n=23, 10) | 87710.8 (18699.28) | 0.7 (44.02)
  AB1-40, Day 240 (n=23, 9) | 20665.6 (7132.91) | -6.2 (35.63)

7. Secondary Outcome: Number of Participants With Brain Structural Magnetic Resonance Imaging (sMRI) Abnormalities
Description: Brain sMRI abnormalities included cerebral edema and total infarcts (including cortical infarcts, white matter infarcts, and subcortical gray matter infarcts). "Total infarcts" is the total number of participants with at least 1 type of infarct.
Time Frame: Baseline/Screening, Day 15, Day 45, Day 90,
Population: All 36 participants who received study treatment were analyzed for this endpoint.
Measure: Number; unit: participants
Arm/Group | PF-04360365 | Placebo
Number analyzed (Participants) | 24 | 12
participants
  Cerebral edema, Screening | 0 | 1
  Cerebral edema, Day 15 | 0 | 1
  Cerebral edema, Day 45 | 0 | 1
  Cerebral edema, Day 90 | 1 | 1
  Total infarcts, Screening | 5 | 3
  Total infarcts, Day 15 | 5 | 3
  Total infarcts, Day 45 | 5 | 3
  Total infarcts, Day 90 | 5 | 3
  Cortical infarcts, Screening | 0 | 0
  Cortical infarcts, Day 15 | 0 | 0
  Cortical infarcts, Day 45 | 0 | 0
  Cortical infarcts, Day 90 | 0 | 0
  White matter infarcts, Screening | 3 | 2
  White matter infarcts, Day 15 | 3 | 2
  White matter infarcts, Day 45 | 3 | 2
  White matter infarcts, Day 90 | 3 | 2
  Subcortical gray matter infarcts, Screening | 3 | 1
  Subcortical gray matter infarcts, Day 15 | 3 | 1
  Subcortical gray matter infarcts, Day 45 | 3 | 1
  Subcortical gray matter infarcts, Day 90 | 3 | 1

8. Secondary Outcome: Mean Montreal Cognitive Assessment (MoCA) Total Score Over Time
Description: The Montreal Cognitive Assessment (MoCA) was used as a safety outcome measure to assess any changes in cognition. The MoCA is a 1-page 30-point test administered in approximately 10 minutes. The MoCA assessed short term memory, visuospatial abilities, multiple aspects of executive functions, attention, concentration, working memory, and language, as well as orientation to time and place. The total scale ranges from 0 to 30, with lower numbers indicating lower cognition performance.
Time Frame: Screening; Days 0, 1, 30, 60, 90, and 240
Population: All 36 participants who received study treatment were included in the analysis. On Day 240, the number of evaluable participants in the placebo group was 11 instead of 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-04360365 | Placebo
Number analyzed (Participants) | 24 | 12
units on a scale
  Screening | 25.4 (4.24) | 25.9 (1.73)
  Day 0 | 25.5 (3.41) | 25.9 (3.34)
  Day 1 | 25.1 (3.10) | 25.8 (2.73)
  Day 30 | 27.0 (2.46) | 26.8 (2.53)
  Day 60 | 26.6 (3.12) | 26.8 (3.33)
  Day 90 | 26.0 (3.46) | 26.7 (3.14)
  Day 240 | 26.1 (3.43) | 26.5 (2.73)

9. Secondary Outcome: Number of Participants With All Causality and Treatment-related Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Discontinuations Due to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. AEs comprised both SAEs and non-SAEs. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent adverse events (TEAEs) were defined as newly occurring AEs or those worsening after first dose.
Time Frame: Baseline up to Day 240
Population: All 36 participants who received study drug were included in the AE summarization/analysis.
Measure: Number; unit: participants
Arm/Group | PF-04360365 | Placebo
Number analyzed (Participants) | 24 | 12
participants
  All causality TEAEs | 16 | 8
  Treatment-related TEAEs | 2 | 2
  All causality SAEs | 2 | 2
  Treatment-related SAEs | 0 | 1
  All causality severe TEAEs | 2 | 2
  Treatment-related severe TEAEs | 0 | 1
  Discontinued due to all causality TEAEs | 0 | 0

10. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Number of participants with laboratory test abnormalities without regard to baseline abnormality. Laboratory test parameters included hematology, liver function (including Hy's Law Criteria), renal function, electrolytes, clinical chemistry, and urinalysis (dipstick and microscopy).
Time Frame: Baseline up to Day 240
Population: All 36 participants who received study drug were included in the analysis.
Measure: Number; unit: participants
Arm/Group | PF-04360365 | Placebo
Number analyzed (Participants) | 24 | 12
participants | 14 | 10

11. Secondary Outcome: Number of Participants With Vital Signs Values Meeting Categorical Summarization Criteria
Description: Categorical summarization criteria in vital signs included: supine systolic blood pressure (SBP) of less than (<)90 millimeters of mercury (mm Hg) or more than (>) 160 mm Hg; supine diastolic blood pressure (DBP) <50 mm Hg or >100 mm Hg; supine pulse rate of <60 beats per minute (bpm) or >100 bpm; maximum changes (increase or decrease) from baseline in supine SBP of >=20 mm Hg; maximum increase from baseline in supine DBP of >=20 mm Hg; and maximum decrease from baseline in supine DBP of >=10 mm Hg.
Time Frame: Baseline up to Day 240
Population: All 36 participants who received study drug were included in the analysis.
Measure: Number; unit: participants
Arm/Group | PF-04360365 | Placebo
Number analyzed (Participants) | 24 | 12
participants
  Supine SBP <90 mm Hg | 1 | 0
  Supine SBP >160 mm Hg | 2 | 2
  Supine DBP <50 mm Hg | 1 | 0
  Supine DBP >100 mm Hg | 0 | 1
  Supine pulse rate <60 bpm | 16 | 7
  Supine pulse rate >100 bpm | 0 | 1
  Increase from baseline in supine SBP >=20 mm Hg | 6 | 4
  Increase from baseline in supine DBP >=20 mm Hg | 1 | 1
  Decrease from baseline in supine SBP >=20 mm Hg | 9 | 6
  Decrease from baseline in supine DBP >=10 mm Hg | 13 | 5

12. Secondary Outcome: Overall Number of Participants With Positive Responses to Questions on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS assessed whether participant responded "yes" to the following: completed suicide, suicide attempt, preparatory acts toward imminent suicidal behavior, suicidal ideation, self-injurious behavior with no suicidal intent.
Time Frame: Baseline up to Day 240
Population: All 36 participants who received study drug were included in the analysis.
Measure: Number; unit: participants
Arm/Group | PF-04360365 | Placebo
Number analyzed (Participants) | 24 | 12
participants
  Completed suicide | 0 | 0
  Suicide attempt | 0 | 0
  Preparatory acts to imminent suicidal behaviour | 0 | 0
  Self-injurious behaviour, no suicidal intent | 1 | 0

13. Secondary Outcome: Number of Participants With Significant Changes From Baseline in Physical Examination at Final Visit
Description: A complete physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, skeletal, and neurological systems.
Time Frame: Baseline up to Final Visit (Day 240)
Population: All 36 participants who received study drug were included in the analysis.
Measure: Number; unit: participants
Arm/Group | PF-04360365 | Placebo
Number analyzed (Participants) | 24 | 12
participants | 0 | 0

14. Secondary Outcome: Number of Participants With Significant Changes in Neurological Examination Results
Description: A complete/full neurological examination included assessment of the cranial nerves; muscle strength, tone, cortical drift, abnormal movements; deep tendon reflexes; sensory exam, coordination, gait and station.
Time Frame: Baseline up till Day 240
Population: All 36 participants who received study drug were included in the analysis.
Measure: Number; unit: participants
Arm/Group | PF-04360365 | Placebo
Number analyzed (Participants) | 24 | 12
participants | 2 | 1

15. Secondary Outcome: Number of Participants With Anti-PF-04360365 Antibodies
Description: Blood samples were collected from participants who received active treatment to assess for presence/absence of anti-PF-04360365 antibodies.
Time Frame: Day 1 up to Day 240
Population: All 24 participants who received PF-04360365 were included in this analysis.
Measure: Number; unit: participants
Arm/Group | PF-04360365
Number analyzed (Participants) | 24
participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious AEs (SAEs) monitoring started from screening through and including 28 calendar days after the last administration of the investigational product.
Description: All treated participants were analyzed for AEs. The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and a nonserious event during the study.
Arm/Group | PF-04360365 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/24 | 2/12
Other Adverse Events (participants affected / at risk) | 16/24 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04360365 (N=24) | Placebo (N=12)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Migraine with aura (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04360365 (N=24) | Placebo (N=12)
Palpitations (Cardiac disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Cerebellar syndrome (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Coordination abnormal (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Superficial siderosis of central nervous system (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Emotional disorder (Psychiatric disorders) | 1 | 0
Testicular cyst (Reproductive system and breast disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.